CLINICAL TRIAL: NCT06617351
Title: The Effect of Melatonin Supplementation on Immune Cell Responses and Functional Recovery Following Acute Resistance Exercise
Brief Title: This Repeated Measures Parallel-group Investigation Will Examine the Influence of Short-term Melatonin Supplementation (5mg, 3 x Day for 72 Hours) on Cellular Responses, Functional Performance and Recovery Following an Acute Bout of Dynamic Resistance Exercise in Resistance Trained Men and Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Adam Wells, Associate Professor of Kinesiology, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00006674
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cell Migration; Cell Invasion; Exercise Recovery
Keywords: melatonin; exercise recovery
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Participants will receive Melatonin (5mg, 3 times daily with breakfast, lunch and dinner) beginning 24 hours before and ending 48 hours following an acute bout of dynamic high-intensity resistance exercise. On the day of the exercise bout, participants will ingest a single dose of Melatonin prior to arriving at the lab and following all testing procedures.
  Melatonin formula: 7.5 kCal, 2 g Carbohydrate, 1.5 g total sugars, 7.5 mg sodium, 5 mg melatonin.
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Participants will receive Placebo (3 times daily with breakfast, lunch and dinner) beginning 24 hours before and ending 48 hours following an acute bout of dynamic high-intensity resistance exercise. On the day of the exercise bout, participants will ingest a single dose of the placebo prior to arriving at the lab and following all testing procedures.
  Placebo formula: 12.5 kCal, 3g Carbohydrate, 1.875 g total sugars, 1.25 mg sodium.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Gummy - 7.5 kilocalories (kCal), 2 g Carbohydrate, 1.5 g total sugars, 7.5 mg sodium, 5 mg melatonin.
  Arms: Melatonin
Dietary Supplement: Placebo — Gummy - 12.5 kilocalories (kCal), 3g Carbohydrate, 1.875 g total sugars, 1.25 mg sodium.
  Arms: Placebo

SUMMARY:
Oral Melatonin is a commercially available product available alone and as a constituent in a number of supplements. Previous research suggests that short-term supplementation with oral melatonin may amplify the recovery response to damaging resistance exercise via modulation of subsequent immune and inflammatory responses. However the effects of oral melatonin on neutrophil and monocyte invasion/migration, a critical step in the resolution of skeletal muscle tissue homeostasis, has not been examined. An oral melatonin supplement (5mg) will be provided three times daily beginning 24-hours before and ending 48-hours after an acute bout of damaging resistance exercise (total 15mg/day for 3 days).

Goals:

1. To investigate the effect of melatonin on systemic and cellular responses following an acute bout of damaging resistance exercise.
2. To investigate the effect of melatonin on measures of functional performance before and during recovery from an acute bout of damaging resistance exercise.

DETAILED DESCRIPTION:
Resistance exercise of sufficient intensity can result in localized damage to skeletal muscle tissue. The resolution of tissue homeostasis following damaging exercise is mediated largely by neutrophils and monocytes of the innate immune system (1). Neutrophils and monocytes originate in the systemic circulation and infiltrate the damaged tissue following activation and migration in response to damage associated molecular cues. These cells are reported to execute a number of processes fundamental to recovery, including the phagocytosis of opsonized cellular debris (2), and secretion of mitogenic factors that stimulate both the proliferation and differentiation of myogenic precursor cells (3). Disruption of this cellular response has been shown to lead to impaired muscle regeneration, and a subsequent deficit in muscle fiber size (4). Accordingly, a successful innate immune response is paramount for optimal tissue regeneration.

Several supplements have been introduced to the market with purported claims of enhanced recovery from exercise. One potential mechanism for enhanced recovery is through augmentation of the immune response, which may allow for a more pronounced stimulus to enhance repair (1). Previous research suggests that short-term supplementation with melatonin, an endogenously produced indoleamine, may amplify the recovery response. Melatonin receptors are expressed on most immune cell types, including monocytes, neutrophils, and Th1 lymphocytes (5). Melatonin has previously been shown to activate monocytes (6), and treatment with melatonin has been shown to upregulate the recruitment of human monocytes through interaction with the melatonin receptor (MLTr) in vitro. Melatonin has also been shown to alter cytokine production and increase the production of cells of both the innate and adaptive immune system (7). Binding of melatonin to MLTr's expressed on immune cells may modulate recruitment of these cells to damaged tissue, which may in turn regulate the ensuing recovery response. Theoretically, this could reduce recovery time following damaging exercise, improving quality of training and potentially allow for enhanced performance over time (8,9,10). Nevertheless, the effect of short-term melatonin supplementation on innate immune cell and inflammatory responses during recovery from resistance exercise has not been examined.

Goals:

1. To assess systemic and cellular responses to an acute bout of resistance exercise between participants ingesting melatonin versus placebo, including creatine kinase (CK), complete blood counts (CBC), serum interleukin-8 (IL-8), serum monocyte chemoattractant protein-1 (MCP-1), serum melatonin, serum C-reactive protein (CRP), cell receptor expression (monocytes: activated CD11b, CCR2, MLTr1A; neutrophils: activated CD11b. CXCR2, MLTr1A), and neutrophil/monocyte invasion/migration dynamics (cell index, CI).
2. To assess functional measures of recovery following an acute bout of resistance exercise between participants ingesting melatonin versus placebo, including subjective sleep quality/duration, fatigue, soreness and stress (Hooper Questionnaire), perceived Recovery (Perceived Recovery Status Scale, PRSS), active range of motion (AROM), pain pressure threshold (PPT), countermovement jump (CMJ), squat maximal voluntary isometric contraction (MVIC), and objective sleep and physical activity (Accelerometry).

Method:

Randomized, double-blind, placebo controlled parallel-groups trial comparing the effect of supplementation with Melatonin versus Placebo on systemic and cellular responses and functional recovery from damaging resistance exercise.

Melatonin or placebo supplementation (randomly assigned) will occur over a period of 3 days beginning 24-hours prior to completion of an acute bout of damaging resistance exercise through a 48-hours post-exercise recovery period.

Objective sleep and physical activity (accelerometry) will be assessed 24-hours before (-24H), 24-hours Post (24H) and 48-Hours (48H) post-exercise. Diet (carbohydrates, fats, proteins, total calories and micronutrients) will be assessed at Pre (0), 24H and 48H post-exercise. CBC, CK, IL-8, MCP-1, CRP, Hooper, PRSS, AROM, PPT, CMJ, MVIC and melatonin will be assessed at Pre (0) immediately- post (IP) 4-hours post (4H), 24H and 48H post-exercise. Neutrophil cell index will be assessed at Pre (0), 4H and 24H post-exercise. Monocyte cell index (CI) will be assessed at Pre (0), 24H and 48H post-exercise. Neutrophil cell receptor expression will be assessed at Pre (0), 4H and 24H. Monocyte receptor expression will be assessed at Pre (0), 24H and 48H.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-40 years old.
* Healthy and ready for physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q+) and Medical History Questionnaire (MHQ).
* Active resistance training for a minimum of 6 months as defined by 3 resistance training sessions (muscle strengthening activities such as free weights, weight machines, or calisthenics, etc.) per week with at least one lower body session as determined by the training history questionnaire.
* Premenopausal, with an identifiable onset of menses (early follicular phase) as determined by the menstrual status questionnaire (female participants only)..
* Not currently pregnant and no intention to become pregnant for the duration of participation (female participants only).
* Currently free from and willing to abstain from dietary supplements that are viewed by study investigators to confound the outcomes of the study (e.g., creatine, beta-alanine) for the duration of the study. Participants currently using supplements will be permitted to enroll in the study following a 4-week washout period of these supplements.
* Willing to adhere to all pre-testing visit instructions including abstaining from exercise for the duration of the study and abstaining from alcohol for 24 hours prior to visit 2 as well as for 24 hours before visit 3 until completion of the study.
* Currently be consuming ≤ 300mg caffeine per day on average and willing to keep caffeine intake consistent throughout the duration of the study. Participants must also be willing to abstain from caffeine intake for 12 hours prior to visits 3, 4 and 5 and not consume caffeine the morning of these visits.
* Free from previous or current lower body injuries that are viewed by the investigators to potentially limit ability of the participant to perform the exercise intervention or functional assessments.
* Not regularly taking any type of prescription or over-the-counter medication which might affect the assessments, or having any chronic illnesses, which require medical care.
* Considered by the study investigators to have a high likelihood of successful venipuncture following an initial examination of the participants antecubital fossa by a certified phlebotomist and verbal discussion of the participants blood draw history (including history of unsuccessful venipunctures, known issues with the locating/palpating of veins in the antecubital fossa by a phlebotomist, and whether these difficulties are more apparent on one arm compared to the other).

Exclusion Criteria:

* Individual does not agree to participate in this study.
* Individual does not meet inclusion criteria to participate in the study protocols as determined via the PAR-Q+, medical history questionnaire, training history questionnaire, and/or the caffeine consumption questionnaire.
* Currently taking melatonin
* Regularly taking any type of prescription or over-the-counter medication which might affect the assessments, or having any chronic illnesses, which require medical care.
* Not currently meeting requirements for resistance trained status.
* Current known pregnancy or intent to become pregnant during the study period.
* Not regularly having periods or amenorrheic, as determined by Menstrual Status Questionnaire (MSQ).
* Currently taking any performance-enhancing drug (determined from health and activity questionnaire).
* Currently taking a nutritional supplement viewed by the research team to confound the outcomes of the study and not willing to abstain from taking the supplement during the course of the study or not willing to undergo a 4-week wash-out period prior to participating if required.
* Evaluated as having a low likelihood of successful venipuncture by a certified phlebotomist.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Sleep Duration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about sleep duration the previous night using the Hooper Questionnaire administered via pen and paper. Response is rated on a seven-point Likert scale with the following responses:
  * 10+
  * 9-10
  * 8-9
  * 8
  * 7-8
  * 5-7
  * 5 or less
Subjective Sleep Quality | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about their sleep quality the previous night using the Hooper Questionnaire administered via pen and paper. Response is rated on a seven-point Likert scale with the following responses:
  * Outstanding
  * Very good
  * Good
  * Better than normal
  * Worse than normal
  * Disrupted
  * Horrible - No Sleep
Subjective Fatigue | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about their current level of fatigue using the Hooper Questionnaire administered via pen and paper. Response is rated on a seven-point Likert scale with the following responses:
  * No Fatigue
  * Minimal Fatigue
  * Better than normal
  * Normal
  * Worse than normal
  * Very Fatigued
  * Exhausted - Major fatigue
Subjective Muscle Soreness | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about their current level of muscle soreness using the Hooper Questionnaire administered via pen and paper. Response is rated on a seven-point Likert scale with the following responses:
  * No Soreness
  * Very little soreness
  * Better than normal
  * Normal
  * Worse than normal
  * Very sore/tight
  * Extremely sore/tight
Subjective Mental Stress | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about their current level of mental stress using the Hooper Questionnaire administered via pen and paper. Response is rated on a seven-point Likert scale with the following responses:
  * Feeling great - Very relaxed
  * Feeling Good - Relaxed
  * Better than normal
  * Normal
  * Worse than normal
  * Stressed
  * Very Stressed
Perceived Recovery Status | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Participants provide information about their perceived recovery status using the Perceived Recovery Status Scale (PRSS). Response is rated on a scale ranging from 0 (very poorly recovered/extremely tired) to 10 (very well recovered/highly energetic). Each response also corresponds to a broader performance categorization with values indicating expectations of either declined performance, similar performance, or improved performance relative to subsequent time points.
Active Range of Motion (AROM) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed in both lower limbs via handheld goniometer while participant is supine. Average of two measures on each limb is used to determine AROM.
Pain Pressure Threshold (PPT) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed in dominant lower limb via manual algometer while participant is supine. PPT is defined as the point at which the pressure applied via the algometer becomes uncomfortable, as verbally indicated by the participant. PPT is measured in triplicate with 10 seconds of rest between measurements. Average of the three measures is used to determine PPT.
Peak Jump Height | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Peak Jump height is the highest jump height across 3 jumps separated by 30 seconds.
Mean Jump Height | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Mean Jump height is the average jump height across 3 jumps separated by 30 seconds.
Peak Jump Force | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Peak force is the highest force achieved across 3 jumps separated by 30 seconds.
Mean Jump Force | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Mean Jump force is the average jump force across 3 jumps separated by 30 seconds.
Peak Braking Force | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Peak braking force is the highest braking force achieved across 3 jumps separated by 30 seconds.
Mean Braking Force | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Mean braking force is the average braking force across 3 jumps separated by 30 seconds.
Peak Braking Rate of Force Development (RFD) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Peak braking rate of force development force is the peak braking RFD force achieved across 3 jumps separated by 30 seconds.
Mean Braking Rate of Force Development (RFD) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Mean braking rate of force development is the average braking RFD force across 3 jumps separated by 30 seconds.
Mean Reactive Strength Index (RSI) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Defined as the time taken to complete the flight phase divided by the total time taken from the initiation of movement to the instant of take-off. Mean RSI is the average RSI across 3 jumps separated by 30 seconds.
Peak Reactive Strength Index (RSI) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via counter movement jump performed using portable force plate system. Defined as the time taken to complete the flight phase divided by the total time taken from the initiation of movement to the instant of take-off. Peak RSI is the peak RSI achieved across 3 jumps separated by 30 seconds.
Squat Maximal Voluntary Isometric Contraction (MVIC) Force | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via isometric squat contraction using portable force plate system and isometric squat rack with fixed bar. Participants will complete three 5-second isometric contractions with one minute of rest between contractions. The highest force achieved during the three contractions will be recorded as Squat MVIC force.
Squat Maximal Voluntary Isometric Contraction (MVIC) Rate of Force Development (RFD) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Determined via isometric squat contraction using portable force plate system and isometric squat rack with fixed bar. Participants will complete three 5-second isometric contractions with one minute of rest between contractions. Rate of force development (RFD), dictated by the onset of muscular contraction, will be recorded at 0-300ms for the contraction with the highest peak force.
Objective Sleep Quality | -24 hours before (-24H), 24-hours Post (24H), 48-hours Post (48H)
  Assessed using an ActiGraph GT9X Link accelerometer. Participants will wear the accelerometer and beginning 24 hours before the resistance exercise protocol through 48-hours post-exercise. Number of minutes that participants are asleep, and the number of times their sleep is disrupted will be assessed.
Physical Activity | -24 hours before (-24H), 24-hours Post (24H), 48-hours Post (48H)
  Assessed using an ActiGraph GT9X Link accelerometer. Participants will wear the accelerometer and beginning 24 hours before the resistance exercise protocol through 48-hours post-exercise. Minutes per day that participants engage in low, moderate, and high intensity physical activity will be assessed.
Hematocrit | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Hemoglobin | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Mean corpuscular volume (MCV) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Mean corpuscular hemoglobin (MCH) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Mean corpuscular hemoglobin concentration (MCHC) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Total white blood cell count (WBC) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Total red blood cell count (RBC) | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Lymphocyte Count | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Monocyte Count | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Granulocyte Count | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Platelet Count | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via Automated Hematology Analyzer
Serum Creatine Kinase (CK) concentration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Marker of muscle damage. Assessed via assay and microplate reader
Serum Melatonin concentration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via assay and microplate reader
Serum C-reactive protein (CRP) concentration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via assay and microplate reader
Serum Interleukin-8 (IL-8) concentration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via assay and microplate reader
Serum Monocyte Chemoattractant Protein-1 (MCP-1) concentration | Pre (0), Immediately-post (IP), 4-hours Post (4H), 24-hours post (24H), 48-hours post (48H)
  Assessed via assay and microplate reader
Monocyte Cell Index (CI) | Pre (0), 24-hours post (24H), 48-hours post (48H)
  Assessed via Real Time Cell Analysis (RTCA) assay
Neutrophil Cell Index (CI) | Pre (0), 4-Hours Post (4H), 24-hours post (24H)
  Assessed via Real Time Cell Analysis (RTCA) assay
Monocyte C-C chemokine receptor 2 (CCR2) expression | Pre (0), 24-hours post (24H), 48-hours post (48H)
  Assessed via flow cytometry
Monocyte Macrophage-1 antigen (Integrin CD11b) expression | Pre (0), 24-hours post (24H), 48-hours post (48H)
  Assessed via flow cytometry
Monocyte Melatonin Receptor 1A (MLTr1A) expression | Pre (0), 24-hours post (24H), 48-hours post (48H)
  Assessed via flow cytometry
Neutrophil Receptor 1A (MLTr1A) expression | Pre (0), 4-Hours Post (4H), 24-hours post (24H)
  Assessed via flow cytometry
Neutrophil Macrophage-1 antigen (Integrin CD11b) expression | Pre (0), 4-Hours Post (4H), 24-hours post (24H)
  Assessed via flow cytometry
Neutrophil Interleukin-8 receptor (CXCR2) expression | Pre (0), 4-Hours Post (4H), 24-hours post (24H)
  Assessed via flow cytometry
Diet - Daily Protein | Pre (0), 24-hours Post (24H), 48-hours Post (48H)
  Assessed via Automated Self-Administered 24hr Dietary Recall (ASA24).
Diet - Daily Carbohydrate | Pre (0), 24-hours Post (24H), 48-hours Post (48H)
  Assessed via Automated Self-Administered 24hr Dietary Recall (ASA24).
Diet - Daily Fat | Pre (0), 24-hours Post (24H), 48-hours Post (48H)
  Assessed via Automated Self-Administered 24hr Dietary Recall (ASA24).
Diet - Daily Total Calories | Pre (0), 24-hours Post (24H), 48-hours Post (48H)
  Assessed via Automated Self-Administered 24hr Dietary Recall (ASA24).
Diet - Daily Total Micronutrients | Pre (0), 24-hours Post (24H), 48-hours Post (48H)
  Assessed via Automated Self-Administered 24hr Dietary Recall (ASA24). Participants report each eating occasion and the time of consumption during a 24-hour period.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinesiology Research Labs, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wells AJ, Hoffman JR, Jajtner AR, Varanoske AN, Church DD, Gonzalez AM, Townsend JR, Boone CH, Baker KM, Beyer KS, Mangine GT, Oliveira LP, Fukuda DH, Stout JR. The Effect of Post-Resistance Exercise Amino Acids on Plasma MCP-1 and CCR2 Expression. Nutrients. 2016 Jul 2;8(7):409. doi: 10.3390/nu8070409. PMID 27384580
- [Background] Aderem A, Underhill DM. Mechanisms of phagocytosis in macrophages. Annu Rev Immunol. 1999;17:593-623. doi: 10.1146/annurev.immunol.17.1.593. PMID 10358769
- [Background] Chazaud B, Brigitte M, Yacoub-Youssef H, Arnold L, Gherardi R, Sonnet C, Lafuste P, Chretien F. Dual and beneficial roles of macrophages during skeletal muscle regeneration. Exerc Sport Sci Rev. 2009 Jan;37(1):18-22. doi: 10.1097/JES.0b013e318190ebdb. PMID 19098520
- [Background] Arnold L, Henry A, Poron F, Baba-Amer Y, van Rooijen N, Plonquet A, Gherardi RK, Chazaud B. Inflammatory monocytes recruited after skeletal muscle injury switch into antiinflammatory macrophages to support myogenesis. J Exp Med. 2007 May 14;204(5):1057-69. doi: 10.1084/jem.20070075. Epub 2007 May 7. PMID 17485518
- [Background] Pozo D, Garcia-Maurino S, Guerrero JM, Calvo JR. mRNA expression of nuclear receptor RZR/RORalpha, melatonin membrane receptor MT, and hydroxindole-O-methyltransferase in different populations of human immune cells. J Pineal Res. 2004 Aug;37(1):48-54. doi: 10.1111/j.1600-079X.2004.00135.x. PMID 15230868
- [Background] Morrey KM, McLachlan JA, Serkin CD, Bakouche O. Activation of human monocytes by the pineal hormone melatonin. J Immunol. 1994 Sep 15;153(6):2671-80. PMID 8077674
- [Background] Calvo JR, Gonzalez-Yanes C, Maldonado MD. The role of melatonin in the cells of the innate immunity: a review. J Pineal Res. 2013 Sep;55(2):103-20. doi: 10.1111/jpi.12075. Epub 2013 Jul 24. PMID 23889107
- [Background] Maldonado MD, Manfredi M, Ribas-Serna J, Garcia-Moreno H, Calvo JR. Melatonin administrated immediately before an intense exercise reverses oxidative stress, improves immunological defenses and lipid metabolism in football players. Physiol Behav. 2012 Mar 20;105(5):1099-103. doi: 10.1016/j.physbeh.2011.12.015. Epub 2011 Dec 22. PMID 22212240
- [Background] Nassar E, Mulligan C, Taylor L, Kerksick C, Galbreath M, Greenwood M, Kreider R, Willoughby DS. Effects of a single dose of N-Acetyl-5-methoxytryptamine (Melatonin) and resistance exercise on the growth hormone/IGF-1 axis in young males and females. J Int Soc Sports Nutr. 2007 Oct 23;4:14. doi: 10.1186/1550-2783-4-14. PMID 17956623
- [Background] Ochoa JJ, Diaz-Castro J, Kajarabille N, Garcia C, Guisado IM, De Teresa C, Guisado R. Melatonin supplementation ameliorates oxidative stress and inflammatory signaling induced by strenuous exercise in adult human males. J Pineal Res. 2011 Nov;51(4):373-80. doi: 10.1111/j.1600-079X.2011.00899.x. Epub 2011 May 26. PMID 21615492